CLINICAL TRIAL: NCT04353258
Title: Using Behavioral Economic Strategies to Address Obesity in Economically Disadvantaged Adults
Brief Title: Research Intervention to Support Healthy Eating and Exercise
Acronym: RISE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Connecticut (Other)
Collaborators: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Responsible Party: Principal Investigator, Tricia Leahey, Associate Professor, University of Connecticut
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: H19-141; 1R01DK118957 (NIH)
Record Dates: First submitted 2020-04-16; First posted 2020-04-20 (Actual); Results first posted 2026-01-09 (Actual); Last update posted 2026-01-09 (Actual); Status verified 2025-07

CONDITIONS: Obesity
Keywords: weight loss, low income, behavioral economics, contingency management, episodic future thinking, mHealth
MeSH Terms: conditions — Obesity; Weight Loss | interventions — Telemedicine

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Behavioral Economics intervention (BE mHealth) (Experimental): Participants will receive a 12-month behavioral weight loss intervention delivered primarily via mobile phone (mHealth) that includes behavioral economics components.
  Interventions: Behavioral: Behavioral Economics intervention (BE mHealth)
- Standard mHealth intervention (mHealth) (Active Comparator): Participants will receive a 12-month behavioral weight loss intervention delivered primarily via mobile phone (mHealth).
  Interventions: Behavioral: Standard mHealth intervention (mHealth)

INTERVENTIONS:
Behavioral: Behavioral Economics intervention (BE mHealth) — Participants will receive a 12-month behavioral weight loss intervention delivered primarily via mobile phone (mHealth) that includes behavioral economics components.
  Arms: Behavioral Economics intervention (BE mHealth)
Behavioral: Standard mHealth intervention (mHealth) — Participants will receive a 12-month behavioral weight loss intervention delivered primarily via mobile phone (mHealth).
  Arms: Standard mHealth intervention (mHealth)

SUMMARY:
The primary aim of this study is to test the efficacy of a behavioral economics intervention for weight loss in adults from economically disadvantaged backgrounds.

ELIGIBILITY:
Inclusion Criteria:

* Age between 18-75
* BMI between 25-55kg/m2
* All sexes
* All racial/ethnic groups
* Low SES and/or report qualifying for federal, state or local benefits
* Have a smartphone and willing to use for research purposes

Exclusion Criteria:

* <18-75>years of age
* Report being unable to walk 2 blocks without stopping
* Are currently participating in weight loss treatment, have a history of bariatric surgery, or lost ≥5% in the past 6-months
* Are pregnant or plan to become pregnant within 1 year
* Report a heart condition, chest pain during periods of rest or activity, or loss of consciousness on the Physical Activity Readiness Questionnaire
* Report a medical condition that could jeopardize their safety in a weight control program with diet and exercise guidelines
* Have diabetes and are on insulin
* Report a medical condition that could jeopardize their safety in a weight loss program with diet and exercise guidelines
* Report conditions that, in the judgment of the PI, would render them unlikely to follow the protocol (e.g., relocation, dementia, unable to read and write in English)
* Report unable to read and write English

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 195 (Actual)
Dates: Start 2021-09-07 (Actual); Primary Completion 2024-12-17 (Actual); Study Completion 2024-12-17 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Tricia Leahey, PhD, Principal Investigator — University of Connecticut
Locations (1):
- UConn Weight Management Research Lab, Hartford, Connecticut, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Behavioral Economics Intervention (BE mHealth) | Standard mHealth Intervention (mHealth)
Started | 97 | 98
Completed | 83 | 85
Not Completed | 14 | 13

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Behavioral Economics Intervention (BE mHealth) | Standard mHealth Intervention (mHealth) | Total
Number analyzed (Participants) | 97 | 98 | 195
Age, Continuous [Mean (Standard Deviation); unit: years] | 37.6 (12.8) | 42.0 (16.9) | 39.7 (15.1)
Sex/Gender, Customized [Count of Participants; unit: Participants]
  Gender: Female | 84 | 84 | 168
  Gender: Male | 13 | 13 | 26
  Gender: Non-binary | 0 | 1 | 1
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 71 | 77 | 148
  Not Hispanic or Latino | 25 | 21 | 46
  Unknown or Not Reported | 1 | 0 | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 2 | 1 | 3
  Asian | 7 | 3 | 10
  Native Hawaiian or Other Pacific Islander | 1 | 0 | 1
  Black or African American | 33 | 37 | 70
  White | 36 | 47 | 83
  More than one race | 10 | 6 | 16
  Unknown or Not Reported | 8 | 4 | 12
Body Mass Index (BMI; kg/m2) [Mean (Standard Deviation); unit: kg/m2] — Weight was assessed objectively via digital scale; height is based on participant's self-report; BMI was calculated using the formula weight in kg / height in m2.
  kg/m2 | 35.7 (7.1) | 34.7 (6.5) | 35.2 (6.8)

OUTCOME MEASURES:

1. Primary Outcome: Weight
Description: Weight change measured on a digital scale to the nearest 0.1-kilogram
Time Frame: Baseline, 2 month, 6 month, 12 month, 18 months
Population: There was attrition over time during this longitudinal study, such that more participants were lost to follow-up over time.
Measure: Mean (Standard Deviation); unit: kg
Arm/Group | Behavioral Economics Intervention (BE mHealth) | Standard mHealth Intervention (mHealth)
Number analyzed (Participants) | 95 | 97
kg
  Baseline | 98.2 (24.5) | 93.5 (19.1)
  2 month: number analyzed (Participants) | 91 | 90
  2 month | 95.3 (23.9) | 91.6 (19.5)
  6 month: number analyzed (Participants) | 84 | 87
  6 month | 93.9 (23.6) | 90.2 (20.5)
  12 month | 94.9 (24.9) | 89.3 (21.0)
  18 month: number analyzed (Participants) | 65 | 60
  18 month | 94.1 (24.7) | 90.9 (20.7)

ADVERSE EVENTS:
Time Frame: Adverse event data were collected over 12 months.
Arm/Group | Behavioral Economics Intervention (BE mHealth) | Standard mHealth Intervention (mHealth)
All-Cause Mortality (participants affected / at risk) | 0/97 | 0/98
Serious Adverse Events (participants affected / at risk) | 3/97 | 6/98
Other Adverse Events (participants affected / at risk) | 7/97 | 5/98
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Behavioral Economics Intervention (BE mHealth) (N=97) | Standard mHealth Intervention (mHealth) (N=98)
Hospitalization (Respiratory, thoracic and mediastinal disorders) | 2 | 0
Hospitalization (Nervous system disorders) | 1 | 1
Hospitalization (Musculoskeletal and connective tissue disorders) | 0 | 1
Hospitalization (Cardiac disorders) | 0 | 2
Hospitalization (Gastrointestinal disorders) | 0 | 2
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Behavioral Economics Intervention (BE mHealth) (N=97) | Standard mHealth Intervention (mHealth) (N=98)
COVID - long/severe (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 2 (2)
Gall Bladder (Gastrointestinal disorders) | 2 | 0
Break/Bad Sprain (Musculoskeletal and connective tissue disorders) | 1 | 3
Pneumonia (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Back issues (Musculoskeletal and connective tissue disorders) | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2025-12-17): https://cdn.clinicaltrials.gov/large-docs/58/NCT04353258/Prot_SAP_000.pdf